CLINICAL TRIAL: NCT02637765
Title: Effect of a Short Program (8 Week) of Increased Physical Activity on Quality of Life of Sedentary Women With Previous Breast Cancer. A Prospective Randomized Trial.
Brief Title: Life ImproVed by Exercise (LIVE Trial)
Acronym: LIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO 121
Record Dates: First submitted 2015-06-19; First posted 2015-12-22 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Physical Activity; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Usual Physical Activity
- Intervention Group (Experimental): 8-week increased physical activity program
  Interventions: Behavioral: Increased Physical Activity

INTERVENTIONS:
Behavioral: Increased Physical Activity — Patients will receive a program of increased physical activity starting from 5000 steps/day up to 12000 steps/day after 8 weeks and an 8-week recreational program of brisk walking/running (3 times a week).
  Arms: Intervention Group

SUMMARY:
This is a prospective randomized controlled trial in which patients with previous breast cancer will be randomized into two treatment arms:

1. Control Group of Usual Physical Activity
2. Intervention Group of Increased Physical Activity

No specific intervention will be performed In the patients randomized in the control group.

Patients randomized in the Intervention group will receive a program of increased physical activity starting from 5000 steps/day up to 12000 steps/day after 8 weeks. At the same time patients of this group will receive an 8-week recreational program of brisk walking/running (3 times a week).

All the patients enrolled in this trial will receive a pedometer device (Garmin Vìvofit) able to count the number of steps, determine a daily goal of steps, determine the covered distance (in Km), determine daily caloric consumption, and determine the movements during sleep.

DETAILED DESCRIPTION:
In this prospective randomized controlled trial patients with previous breast cancer will be randomized into two treatment arms:

1. Control Group of Usual Physical Activity
2. Intervention Group of Increased Physical Activity

No specific intervention will be performed In the patients randomized in the control group.

Patients randomized in the Intervention Group will receive a program of increased physical activity starting from 5000 steps/day up to 12000 steps/day after 8 weeks. At the same time patients of this group will receive an 8-week recreational program of brisk walking/running (3 times a week).

All the patients enrolled in this trial will receive a pedometer device (Garmin Vìvofit) able to count the number of steps, determine a daily goal of steps, determine the covered distance (in Km), determine daily caloric consumption, and determine the movements during sleep.

Data will be downloaded in a specific application available online (Garmin Connect).

All the patients will receive written information on the potential benefits of physical exercise and better lifestyle.

At baseline, at the end of the study period (8 weeks) and after 1 year patients will be asked to fill out the following questionnaires:

* Funcional Assessment of Cancer Therapy- Breast (FACT-B, 37 items)
* Patient reported symptoms (PRS like International Breast Cancer Study Group form, 19 items)
* Funcional Assessment of Cancer Therapy- Fatigue (FACT-Fatigue, 13 items)
* Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog; 37 items)
* Impact of Event Scale (IES; 22 items)

At baseline, at the end of the study period (8 weeks) patients will be asked to undergo blood draw for serum analysis of insulin, IGF-1, leptin, PCR, cholesterol, triglycerides leucocyte count, T lymphocyte subpopulations (T regulatory and TH17).

The hypothesis of the study is that even a short course of increased physical activity may improve quality of life of non-regular exercisers women with a personal history of breast cancer who completed treatment (endocrine treatment excluded).

ELIGIBILITY:
Inclusion Criteria:

* Women with personal history of breast cancer AND
* Written informed consent AND
* Willing to be randomized to either group AND
* Age 18-70 years
* Treatment (surgery, chemotherapy, radiotherapy, trastuzumab) completed since at least 6 months and up to 3 years (endocrine therapy allowed)
* Non regular exercisers (≤150 minutes per week of moderate-intense exercise).

Exclusion Criteria:

* Diabetes or other insulin metabolic impairment
* General contraindications to regular physical activity participation
* Inability to ambulate
* Plan to relocate far from the study site
* Presence of any severe medical condition such that the patient is not expected to adhere at the planned study protocol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
quality of life | 8 weeks
  questionnaire

SECONDARY OUTCOMES:
self-report questionaire of principal side effects of medical treatments | 8 weeks
patients' self-reported perceptions of their cognitive abilities | 8 weeks
  37 items consisting of 1) patients' perceived cognitive impair- ments, 2) perceived cognitive abilities, 3) noticeability or com- ments from others, and 4) impact of cognitive changes on quality of life
subjective response to a specific traumatic event | 8 weeks
  administration of self-report validated questionnaire
body weight | 8 weeks
  Registration of body weight at baseline and 8 weeks
sleep | 8 weeks
  Registration of movements during sleep (Data registered by the pedometer device)
insulin | 8 weeks
  serum analysis at baseline and 8 weeks
immune function (as determined by Th17 e T regulators) | 8 weeks
  serum analysis at baseline and 8 weeks
IGF-1 | 8 weeks
  serum analysis at baseline and 8 weeks
Leptin | 8 weeks
  serum analysis at baseline and 8 weeks
C Reactive Protein | 8 weeks
  serum analysis at baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oreste D Gentilini, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy